CLINICAL TRIAL: NCT01604642
Title: Role of Activin A (ActA) in the Human Cancer Cachexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ACTICA
Record Dates: First submitted 2012-05-04; First posted 2012-05-24 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer; Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cachectic versus no cachectic patients (Other): blood tests, muscular biopsies
  Interventions: Other: blood tests and muscular biopsies

INTERVENTIONS:
Other: blood tests and muscular biopsies — blood tests and muscular biopsies

SUMMARY:
The goal of the investigators study is to investigate the role of a hormone named Activin A (ActA) in the development of the skeletal muscle atrophy caused by cancer. According to the investigators hypothesis, ActA could be released by the tumor and activate a muscle atrophy gene program. To answer this question, the investigators plan first to compare circulating levels of ActA in cancer patients with and without cachexia. In a second step, the investigators would like to assess whether ActA circulating levels are predictive for the development of cachexia and short survival.

ELIGIBILITY:
Inclusion Criteria:

* 18-year-old or older
* Colorectal or lung cancer demonstrated by histology or cytology
* New diagnosis or new recurrence
* Expected survival more than 3 months
* No previous history of other cancer in the last 5 years
* No pregnancy or lactation
* Signed informed consent

Exclusion Criteria:

* Non-caucasian
* Major digestive malabsorption
* Major depression
* Artificial nutrition
* Height doses of steroids (>1 mg/kg hydrocortisone equivalent)
* Hyperthyroidism
* Other causes of malnutrition
* Expected survival less than 3 months
* Severely impaired walking
* Anticoagulants or antiplatelet therapy
* Disability or medical condition which might prevent the compliance to the protocol
* Any conditions which may prevent the compliance to the protocol
* Performance status ECOG > ou = 4
* Participation to other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Circulating Activin A level | 2 years

SECONDARY OUTCOMES:
Dietary assessment measured by SNAQ score and 3-Day intake | 2 years
Body mass index | 2 years
Mid arm muscle circumference calculated by the triceps skinfold and the mid arm circumference | 2 years
Body composition measured by bioimpedance | 2 years
Muscle strength as measured by grip strength | 2 years
Quality of life as assessed using the QLQ-C30 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Loumaye A, de Barsy M, Nachit M, Lause P, Frateur L, van Maanen A, Trefois P, Gruson D, Thissen JP. Role of Activin A and myostatin in human cancer cachexia. J Clin Endocrinol Metab. 2015 May;100(5):2030-8. doi: 10.1210/jc.2014-4318. Epub 2015 Mar 9. PMID 25751105